CLINICAL TRIAL: NCT02948933
Title: Post-Authorization Safety Study: Cohort Event Monitoring for Dengvaxia®, CYD-TDV Dengue Vaccine
Brief Title: Cohort Event Monitoring for Dengvaxia®, CYD-TDV Dengue Vaccine
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: DNG15; U1111-1143-8608 (Registry Identifier: ICTRP); EUPAS28947 (Registry Identifier: ENCEPP)
Record Dates: First submitted 2016-10-27; First posted 2016-10-31 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Dengue Fever; Dengue Hemorrhagic Fever
Keywords: Dengue Fever; Dengue Hemorrhagic Fever; Dengvaxia®
MeSH Terms: conditions — Dengue; Severe Dengue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to evaluate the safety profile of Dengvaxia® when used in the real-world immunization setting

Primary Objective:

* To measure the incidence of selected adverse events (AEs) and serious AEs (SAEs) occurring over a period of six (6) months after each Dengvaxia® dose administration;
* To quantify the association between Dengvaxia® and each of the selected AEs and SAEs for which a risk window after vaccination can be defined, using estimates of relative risk
* To monitor the occurrence and frequency of hospitalized dengue disease as well as any other SAEs leading to hospitalization or death, including new and previously unrecognized SAEs, following Dengvaxia® administration on a longer term (up to 5 years after the first Dengvaxia® dose administration.

Secondary objectives:

* To identify risk factors for hospitalized dengue disease (severe or not) among subjects vaccinated with Dengvaxia®;
* To describe the frequency of hospitalized dengue disease and/or other SAEs or selected AEs according to the number of Dengvaxia® doses and/or interval between doses.

DETAILED DESCRIPTION:
This is a prospective multi-national non-interventional study that includes two components of Cohort Event Monitoring (i) Short-term safety surveillance with a follow-up of 6 months after each Dengvaxia® dose administration and (ii) a long-term safety surveillance with a follow-up of five years after the first dose.

No vaccine will be provided as part of this study.

Study population will be identified in a convenient sample of sites as representative as possible of vaccination centers in each country. Subjects who received their first dose of Dengvaxia® at participating sites during the recruitment period and who meet the eligibility criteria will be asked to participate. After enrollment, vaccinees will be contacted periodically by telephone, e-mail, or Short Message Service (SMS) during follow-up for the identification of outcomes and Dengvaxia® vaccination status.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who received the first dose of Dengvaxia® across all age groups, even if vaccination was given outside of local specific label indications or recommendations
* Informed consent form (ICF) or Assent form (AF) has been signed and dated by the subject (based on local regulations), and/or ICF has been signed and dated by the parent(s) or another legal acceptable representative (and by an independent witness if required by local regulations)
* Subjects for whom a telephone contact or an e-mail address is available.

Exclusion Criteria:

* None

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study population will be identified in a convenient sample of sites as representative as possible of vaccination centers in each country. Subjects who received their first dose of Dengvaxia® across all age groups at participating sites during the recruitment period and who meet the eligibility criteria will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with selected adverse events leading to a medical consultation, emergency room visit or hospitalization occurring during the short term surveillance period of 6 months after each dose of Dengvaxia® | 6 months post-vaccination
Percentage of subjects hospitalized with dengue disease (regardless of severity and laboratory confirmation of diagnosis) after each dose of Dengvaxia®. | 6 months post-vaccination
Percentage of subjects with any other serious adverse events (SAEs) occurring during the short term surveillance, and SAEs leading to hospitalization or death occurring during the long term surveillance | Up to 5 years post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Ltd.

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com